CLINICAL TRIAL: NCT07060547
Title: Investigating HepQuant DuO Test as a Biomarker in Alcohol-related Liver Disease
Status: Recruiting | Type: Observational
Sponsor: HepQuant, LLC (Industry)
Collaborators: Leland Stanford Junior University (Unknown)
Responsible Party: Sponsor
Other Study IDs: Stanford 78916
Record Dates: First submitted 2025-05-13; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Alcoholic Hepatitis; Alcohol-related Liver Disease
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: HepQuant DuO Test — HepQuant DuO is commercially available in the U.S. as a Laboratory Developed Test (LDT), but it will be used in this study as a nonsignificant risk investigational device to measure change in liver function over time.

SUMMARY:
This is a study to measure liver recovery in patients with recent alcohol-associated liver injury by assessing liver function and physiology using HepQuant DuO. The HepQuant DuO Test is a blood-based test that involves a drink of a natural compound, cholate, and 2 blood samples at 20 and 60 minutes. The study team is collecting clinical and laboratory data to better monitor and treat patients who have been affected by alcohol-associated liver disease. The study has 4 visits at an outpatient clinic at 1, 3, 6, and 12 months. At each of these visits, participants will undergo a HepQuant DuO test and other standard tests. In addition, the study team will ask about a participant's alcohol use, symptoms, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* adult with a clinical diagnosis of liver disease due to alcohol who have acute hepatic decompensation.

adult with a combined clinical diagnosis of alcohol-related liver disease (ALD) and nonalcoholic steatohepatitis (NASH).

Exclusion Criteria:

* Clinical diagnosis of liver disease with an etiology other than alcohol liver disease unless it is a combined clinical diagnosis of ALD and NASH.
* patients with solid organ malignancy.
* patients with other disease affecting the liver including autoimmune, drug-related liver injury, hemochromatosis or Wilson's disease
* pregnancy
* under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Identify patients through an automated report run in electronic medical record and notifications by treating physicians on the hepatology consult service. No recruitment materials (e.g. flyers) will be used as all patients are identified and enrolled as inpatients.
  Potential participants identified during the chart review will be notified that they may be eligible for this research study by their primary inpatient medical team (MD). Patients will be contacted only after the patient's physician has previously notified the potential research participant and obtained approval for such contact.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Change in HepQuant Disease Severity Index (DSI) over time in patients with ALD | From enrollment to 1 year past enrollment
  The objective of use of the HepQuant DuO test in this study is to evaluate how the HepQuant Disease Severity Index (DSI) changes over time in patients with alcohol-related liver disease (ALD) and to define the relationships of change in HepQuant DSI (ΔDSI) to the changes in the standard of care laboratory and imaging tests used for measuring severity of liver disease and clinical outcomes. The HepQuant DSI is a value on a scale of 0 to 50, where 0 indicates no liver disease and 50 indicates severe liver disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Dept. of Medicine -Gastroenterology & Hepatology, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No